CLINICAL TRIAL: NCT02584296
Title: Physical Activity as a Self-Management Approach to Improve Health Outcomes in Acute Myeloid Leukemia
Brief Title: Physical Activity as Self-Management Approach to Improve Health Outcomes in AML
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Massey Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: MCC-15-11061; HM20004012
Record Dates: First submitted 2015-09-28; First posted 2015-10-22 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Leukemia; Myeloid; Monocytic
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual care control (No Intervention): Phase 1 will be observation only, and will be considered a usual care control group, activity at home.
- Biobehavioral self management approach (Experimental): Phase 2 participants will receive the Biobehavioral self management approach (BSMA) intervention aligned with the IMB model; introduced over three days of each five-day consolidation chemotherapy hospital admission.
  Interventions: Behavioral: BSMA

INTERVENTIONS:
Behavioral: BSMA — Biobehavioral self-management approach (BSMA) intervention is aligned with information-motivation-behavioral skills (IMB) model and is guided physical activity (PA). Collects demographic, medical, disease, treatment data, blood specimens and the battery of measures. Includes PA self-assessment, 6 minute walk test(6MWT) and chair squat test (CST) with Physical Therapist (PT); provides PA handouts based on American Cancer Society (ACS) guidelines, discusses known benefits, beliefs and goals of PA (IMB health behavior motivation); assess/discuss perceived barriers to PA. PT or Exercise physiologist (EP) works with subject on various exercises (both strength and aerobic, ~30 minutes; IMB behavioral skills);PT or EP reviews exercises, subject practices, and provides a BSMA program (including strength/aerobic training) for subject to begin upon discharge. Subject keeps journal of PA and wears accelerometer (TAA) to record PA levels. 3-weeks at home study nurse calls subjects each week.
  Other Names: Biobehavioral self management approach
  Arms: Biobehavioral self management approach

SUMMARY:
Physical Activity as a Self-Management Approach to Improve Health Outcomes in Acute Myeloid Leukemia

DETAILED DESCRIPTION:
Guided by the information-motivation-behavioral skills model and using a quasi-experimental cohort control research design, the primary aim of this study is to: Determine the feasibility of the biobehavioral self management approach (BSMA) program involving physical activity (PA) in patients receiving consolidation treatment for AML. The primary feasibility outcomes for this aim will be rates of recruitment, refusal, retention and attrition; in addition investigators will test methods and procedures of the prescribed BSMA PA program, including assessing adherence, participant acceptance and perceived benefit.

ELIGIBILITY:
Inclusion criteria:

* ≥18 years
* diagnosis of AML
* hospitalized for consolidation chemotherapy within 1 day (+/- 2 days)
* read and write in English
* able to stand independently
* not experiencing psychiatric neurological disorders (assessed through clinical team members) that would prevent obtaining consent.

Exclusion criteria:

* currently experiencing psychiatric or neurologic disorders that would prevent their ability to provide consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-03; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Rates of recruitment, refusal, retention, and attrition will be aggregated to determine the feasibility of the BSMA program for patients receiving consolidation treatment for AML. | 3 months
  These aggregated rates will help determine the feasibility of the biobehavioral self-management approach (BSMA) program involving physical activity (PA) in patients receiving consolidation treatment for acute myeloid leukemia (AML). The primary aim of this study rates of recruitment, refusal, retention, and attrition in the BSMA program for patients receiving consolidation treatment for AML will be reported rates of recruitment (number enrolled, refused), retention, and adherence (trends in exercise capacity as measured by 6minute walk test, strength test and chair to stand test; completed physical activity log; and accelerometer data).

CONTACTS AND LOCATIONS:
Overall Officials: Tara Albrecht, PhD, ACNP-BC, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia, United States